CLINICAL TRIAL: NCT05369468
Title: Efficacy of Adding Dexmedetomidine to Bupivacaine in Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia After Laparoscopic Cholecystectomy: A Prospective Randomized Trial
Brief Title: Dexmetomidine With Erector Spinae Plane Block in Cholecystectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Wafaa Madhy Atia Abdelwahed, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 35225/1/22
Record Dates: First submitted 2022-04-23; First posted 2022-05-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Dexmedtomidine in Erector Spinae Block for Laparscopic Cholecystectomy
Keywords: dexmedtomidine-erector spinae block-cholecystectomy
MeSH Terms: interventions — Dexmedetomidine; Adjuvants, Pharmaceutic; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: both investigator and outcome assessor do not know in which group is the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Placebo Comparator): Group 1: will receive bilateral ESP block with injection of 20 ml of 0.25% Bupivacaine in each site of injection .
  Interventions: Drug: Bupivacain only
- group 2 (Experimental): Group 2: will receive bilateral ESP block with injection of 18ml of 0.25% Bupivacaine plus 2ml dexmedetomidine 0.5 ug /kg in each site of injection .
  Interventions: Drug: dexmedetomidine as adjuvant with bupivacaine

INTERVENTIONS:
Drug: dexmedetomidine as adjuvant with bupivacaine — to assess efficacy of adding dexmedetomidine as adjuvant with bupivacaine in ultrasound-guided erector spinae plane block in patient undergoing laporoscopic cholecystectomy. primary outcome was the total amount of morphine consumption in the first 24-hour postoperative, and the secondary outcomes were the time of first rescue analgesia ,pain score, and safety.
  Arms: group 2
Drug: Bupivacain only — to assess efficacy of bupivacain alone in ultrasound-guided erector spinae plane block in patient undergoing laporoscopic cholecystectomy. primary outcome was the total amount of morphine consumption in the first 24-hour postoperative, and the secondary outcomes were the time of first rescue analgesia ,pain score, and safety.
  Arms: group 1

SUMMARY:
Sixty patients scheduled for elective laparoscopic cholecystectomy will be randomly assigned using sealed envelope into two equal groups (30 patients each).

Group 1: will receive bilateral ESP block with injection of 20 ml of 0.25% Bupivacaine in each site of injection .

Group 2: will receive bilateral ESP block with injection of 18ml of 0.25% Bupivacaine plus 2ml dexmedetomidine 0.5 ug /kg in each site of injection .

DETAILED DESCRIPTION:
This prospective randomized study will be carried out in general surgery Department within 6 months from January 2022 to June 2022 on the 60 patients scheduled for elective laparoscopic cholecystectomy . A written informed consent will be obtained from the patients. Every patient will receive an explanation to the purpose of the study and will have a secret code number and the photos applied only to the part of the body linked to the research to ensure privacy to participants and confidentiality of data.

Research results will be only used for scientific purposes. Procedures will be approved by both the Institutional and the Regional ethical committees.

The risk that may occur is minimal, inadequate analgesia and this risk will be overcome by tramadol 50 mg intravenously STAT dose. Any unexpected risk appears during the course of the research will be cleared to the participants and ethical committee on time and proper measures will be taken to overcome or minimize these risks.

The research end point when reach desired lower pain score postoperative without occurance of any complication as heamodynamic instability.

. Preanesthetic checkup and routine investigations, such as complete blood count test, liver &kidney function test and coagulation profile, will be done. Patients will be kept fasting for 8 h.

On arrival in the operative room, standard monitoring equipment will be attached (electrocardiogram, pulse oximeter, and noninvasive blood pressure) and baseline vital parameters such as heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), respiratory rate (RR), and oxygen saturation (SpO2) will be noted just before induction of anesthesia. Peripheral venous access will be obtained IV crystalloid at rate 10 ml\kg will be infused.

Technique of ultrasound guided Erector spine plane block:

The pa¬tient will be placed in sitting position and the ultrasound-guided ESP block was performed bilaterally at the (T7) level. A 23 G spinal needle was inserted with the bevel in cephalo- caudal direction .

Sixty patients will be randomly assigned using sealed envelope into two equal groups (30 patients each).

Group 1: will receive bilateral ESP block with injection of 20 ml of 0.25% Bupivacaine in each site of injection .

Group 2: will receive bilateral ESP block with injection of 18ml of 0.25% Bupivacaine plus 2ml dexmedetomidine 0.5 ug /kg in each site of injection .

Anesthesia will be induced with injection of propofol 2 mg/kg, and fentanyl 1ug/kg intravenous (I.V) Endotracheal intubation will be facilitated with injection rocuronium bromide 0.9 mg/kg IV. Anesthesia will be maintained with in O2 with sevoflurane 2% to maintained BIS 40-60. Neuromuscular relaxation will be maintained with injection rocuronium top ups of 0.3 mg i.v every hour.

The lungs will be mechanically ventilated to keep end-tidalCO2 within normal range and residual neuromuscular block will be reversed with injection neostigmine (0.05 mg/kg) and injection atropine (0.01 mg/kg). The patients will be extubated when respiration deemed sufficient. The patients will be transferred to recovery room. In the post anesthesia care unit(PACU), they will be monitored for any evidence of complications or adverse events and discharged when aldert score ≥ 9.

ELIGIBILITY:
* Patients undergoing elective laparoscopic cholecystectomy
* aged 18-65 years old
* ASA physical status I or II.

Exclusion Criteria:

* patients who refuse to give written informed consent

  * sever respiratory or cardiac disorder
  * coagulopathy
  * local infection at injection site
  * spine or chest wall deformity
  * patients with known allergy to the drugs used

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption | first 24 hours
  the total amount of morphine consumption in the first 24-hour postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
the result will be shared only after completion of the study and publication